CLINICAL TRIAL: NCT03785951
Title: Impact of Whey and Leucine on Glycaemia in Adults Without Diabetes But With Moderately Raised HbA1c
Brief Title: Impact of Whey and Leucine on Glycaemia in Adults Without Diabetes
Acronym: Whey2Glo
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Reading (Other)
Collaborators: Barnham Benevolent Foundation (Unknown); Jason and Daphne Mermikides Charitable Trust (Unknown)
Responsible Party: Principal Investigator, Julie Lovegrove, Professor, University of Reading
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Prevention
Other Study IDs: 17/56
Record Dates: First submitted 2018-12-14; First posted 2018-12-24 (Actual); Last update posted 2018-12-24 (Actual); Status verified 2018-12

CONDITIONS: Pre Diabetes
Keywords: HbA1c; whey; postprandial glycaemia; cardiometabolic; vascular; leucine; branched chain amino acids (BCAA); glucose control; Milk protein
MeSH Terms: conditions — Glucose Intolerance | interventions — Leucine

STUDY DESIGN:
Intervention Model Description: Double-blind, randomised, controlled, 3-way, cross-over study
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Coded protein products will be used.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Whey Protein Isolate (Experimental): Subjects are asked to supplement their habitual diet with 56 g of whey protein isolate a day for 8 weeks
  Interventions: Dietary Supplement: Whey Protein Isolate; Dietary Supplement: Wheat Protein; Dietary Supplement: Wheat Protein with Leucine
- Wheat Protein (Experimental): Subjects are asked to supplement their habitual diet with 56 g of wheat protein a day for 8 weeks
  Interventions: Dietary Supplement: Whey Protein Isolate; Dietary Supplement: Wheat Protein; Dietary Supplement: Wheat Protein with Leucine
- Wheat protein with leucine (Experimental): Subjects are asked to supplement their habitual diet with 56 g of wheat protein with leucine a day for 8 weeks
  Interventions: Dietary Supplement: Whey Protein Isolate; Dietary Supplement: Wheat Protein; Dietary Supplement: Wheat Protein with Leucine

INTERVENTIONS:
Dietary Supplement: Whey Protein Isolate — Whey protein product isolated from whole milk. 79% Protein with minimal carbohydrate and fat.
  50 grams of total supplemental protein/amino acids from whey protein powder consumed in two 25g (total protein/amino acids) nutrition shakes twice per day for 8 weeks in the form of a nutritional shake.
Dietary Supplement: Wheat Protein — Enzymatically hydrolysed wheat protein containing wheat peptides. 75% Protein with minimal carbohydrate and fat.
  50 grams of total supplemental protein/amino acids from whet protein peptide powder consumed in two 25g (total protein/amino acids) nutrition shakes twice per day for 8 weeks in the form of a nutritional shake.
Dietary Supplement: Wheat Protein with Leucine — Enzymatically hydrolysed wheat protein containing wheat peptides with and additional 1.4g of L-leucine. 75% Protein with minimal carbohydrate and fat and a L-leucine concentration equal to whey protein isolate.
  50 grams of total supplemental protein/amino acids from wheat protein peptide powder, with added leucine to equal the total content of the whey protein condition, consumed in two 25g (total protein/amino acids) nutrition shakes twice per day for 8 weeks.

SUMMARY:
Higher than average blood sugar (glucose) levels are linked to an increased risk of developing type 2 diabetes. As such, there is interest in identifying dietary factors that could lower blood glucose to help reduce the number of people with this disease. Findings from some human studies indicate that dairy products, especially a milk protein (whey), may help the control of blood glucose levels. However, there is a need for further studies to confirm these findings in individuals without diabetes but with higher than average blood glucose levels.

DETAILED DESCRIPTION:
In the UK, more than 700 people are diagnosed with type 2 diabetes each day. Higher than average (raised) fasting blood sugar (glucose) is a characteristic of those at risk of developing this disease and as a result there is significant interest in dietary factors that could reduce levels of blood glucose, lowering the frequency of type 2 diabetes in the population. Existing scientific evidence suggests an important role of dairy products and especially of whey protein in the control of blood glucose levels. However, there is a need for further studies to confirm these findings in individuals without diabetes but with higher than average blood glucose levels.

Milk contains high quality proteins, of which 80% are caseins and 20% are whey proteins. Whey proteins are a rich source of branched-chain amino acids (such as leucine) which are thought to play an important role in regulating blood glucose control and other aspects of cardiovascular disease development in both healthy and type 2 diabetic subjects. However, very few studies in non-diabetic subjects with moderately raised HbA1c, characteristic of long-term poor glucose control, have been performed to investigate how whey protein affects blood glucose levels in the body especially when consumed over the longer term in the daily diet. Furthermore, data are limited on whether the leucine content of protein plays an important role in controlling blood glucose levels.

Study aims The main aims of this study is to investigate in adults without diabetes but with moderately raised HbA1c (a long- term marker of blood glucose control) whether a protein obtained from milk and dairy products (whey) has a beneficial effect on fasting and day-long blood glucose and insulin levels compared with a plant based protein (such as wheat). The researchers will also determine if leucine, a particular amino acid (building blocks of protein) found in higher levels in whey protein plays an important role in controlling blood glucose levels.

A secondary aim will determine whether the protein interventions influence risk markers for developing heart disease and diabetes including the level of blood lipids, hormones regulating blood sugar levels and blood vessel health.

This study will test the hypothesis that the incorporation of whey protein (total protein dose 50 g/d) in the habitual diet for 8 weeks will result in an improvement in fasting and day-long blood glucose and insulin levels, and other risk markers of heart disease and diabetes compared with wheat protein (total protein dose 50 g/d), and that the addition of leucine to wheat (to match the content found in whey protein) will improve blood glucose control.

Study design This study will be a long term, double-blind, randomised, controlled, three-way, cross-over study, in which the participants will receive the protein supplements (in random order) for 8 weeks each, with a 4 week wash-out period between the different protein treatments. At the beginning and end of each protein intervention, a fasting blood sample will be collected to determine the longer term effects of the assigned protein supplement on fasting glycaemic control, insulin sensitivity, endothelial function and other cardio-metabolic risk markers, as well as non-invasive measures of blood vessel health. At the beginning of each intervention period, a subset of participants will also undergo a day-long test meal investigation to determine the short-term (postprandial) effects of the protein interventions on the study outcome measures in response to standard sequential test meals containing the assigned protein interventions.

ELIGIBILITY:
Inclusion Criteria:

* BMI 20-35 kg/m2
* HbA1c (5.7 - 6.5%) or (38.8 - 47.5 mmol/mol)
* Fasting glucose 5.5-6.9 mmol/l
* Fasting total cholesterol <7.5mmol/l
* Fasting triacylglycerol <4.0 mmol/l
* Not having a milk, gluten or wheat allergy or lactose intolerability
* Not having diabetes (HbA1c < 47 mmol/mol) or < 6.5%
* Not suffering from cardiovascular, renal, gastrointestinal, respiratory, endocrine or liver disease
* Not having hypertension
* Not diagnosed with cancer
* Not having surgery in the previous 6 months
* Not consuming more than the recommended intake of alcohol (>14 unit/wk)
* Not being a blood donor 3 months prior to or during the study.
* Not taking extra protein powder supplements in the previous 2 months
* Not anaemic (Haemoglobin ≥115 g/l for women and ≥ 130 g/l for men)
* Not taking medication for raised blood lipids, high blood pressure or for inflammatory conditions.

Exclusion Criteria:

• Females who are breast-feeding, may be pregnant, or if of child-bearing potential and are not using effective contraceptive precautions

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2018-12 (Estimated); Primary Completion 2020-07 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Change in fasting and day long glucose levels | Before and after each 8 week intervention.
  Blood glucose levels will be measured using a clinical chemistry analyser
Change in fasting and day long insulin levels | Before and after each 8 week intervention.
  Blood insulin levels will be measured using ELISA

SECONDARY OUTCOMES:
Change in vascular reactivity measured by Laser Doppler Imaging with iontophoresis | Before and after each 8 week intervention.
  Fasting and day long measurement of vascular reactivity in the microcirculation.
Change in the total and HDL-cholesterol | Before and after each 8 week intervention
  Fasting total cholesterol and HDL-C will be measured using a clinical chemistry analyser. LDL-C will be calculated using the Friedewald formula
Change in fructosamine | Before and after each 8 week intervention
  Fructosamine will be measured using a clinical chemistry analyser
Change in C-reactive protein | Before and after each 8 week intervention
  C-reactive protein
Change in pulse wave analysis | Before and after each 8 week intervention
  Pulse wave analysis will be measured using the Mobil-O-Graph device
Change in blood pressure | Before and after each 8 week intervention
  Systolic blood pressure, diastolic blood pressure and pulse pressure
Change in cellular adhesion molecule | Before and after each 8 week intervention
  VCAM and ICAM will be measured by Luminex, ICAM, P-selectin and E-selectin
Change in selectins | Before the start of the intervention
  P-selectin and E-selectin will be measured using Luminex
Change in beta-hydroxy butyrate | Before and after each 8 week intervention
  Beta-hydroxy butyrate will be measured using a clinical chemistry analyser as a marker of ketone bodies
Change in insulin sensitivity | Before and after each 8 week intervention
  Glucose and insulin levels will be used to estimate insulin sensitivity using the Homeostatic model assessment calculation
Change in non-esterified fatty acids | Before and after each 8 week intervention
  Non-esterified fatty acids will be measured using a clinical chemistry analyser
Measurement of height | Before the start of the intervention
  Height will be measured using a stadiometer
Change in body weight | Before and after each 8 week intervention
  Body weight will be measured using the Tanita scale
Change in body mass index | Before and after each 8 week intervention
  Body mass index will be calculated from body weight and height measurement
Change in body composition | Before and after each 8 week intervention
  Body composition will be measured using bioelectrical impedance.

OTHER OUTCOMES:
Metabonomics | Before and after each 8 week intervention
  Urinary biomarkers will be measured using NMR

CONTACTS AND LOCATIONS:
Overall Officials: Julie Lovegrove, Professor, Principal Investigator — University of Reading
Locations (1):
- Hugh Sinclair Unit of Human Nutrition, Department of Food and Nutritional Sciences, University of Reading, Reading, Berkshire, United Kingdom

REFERENCES:
- [Background] Pal S, Ellis V, Dhaliwal S. Effects of whey protein isolate on body composition, lipids, insulin and glucose in overweight and obese individuals. Br J Nutr. 2010 Sep;104(5):716-23. doi: 10.1017/S0007114510000991. Epub 2010 Apr 9. PMID 20377924
- [Background] Nilsson M, Stenberg M, Frid AH, Holst JJ, Bjorck IM. Glycemia and insulinemia in healthy subjects after lactose-equivalent meals of milk and other food proteins: the role of plasma amino acids and incretins. Am J Clin Nutr. 2004 Nov;80(5):1246-53. doi: 10.1093/ajcn/80.5.1246. PMID 15531672